CLINICAL TRIAL: NCT05808790
Title: Colorectal Pulmonary Metastases: Pulmonary Metastasectomy Versus Stereotactic Ablative Radiotherapy: a Phase III Multicenter Randomized Controlled Trial
Brief Title: Colorectal Pulmonary Metastases: Pulmonary Metastasectomy Versus Stereotactic Ablative Radiotherapy
Acronym: COPPER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Martijn van Dorp, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABR 82437
Record Dates: First submitted 2023-03-24; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Lung Metastases; Colorectal Cancer Metastatic
Keywords: Colorectal pulmonary metastases; Pulmonary metastasectomy; Stereotactic radiotherapy; Randomized controlled trial; Colorectal cancer metastases
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Multicenter, parallel-arm, phase III randomized controlled trial Patients will be randomized in a 1:1 manner to SABR or minimally invasive metastasectomy for the local treatment of three or less colorectal pulmonary metastases
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive pulmonary metastasectomy (Active Comparator): Minimally invasive parenchymal sparing pulmonary metastasectomy Surgical approach by means of video-assisted thoracic surgery (VATS), robot-assisted (RATS), or uniportal VATS
  Interventions: Procedure: Minimally invasive pulmonary metastasectomy
- Stereotactic ablative radiotherapy (Experimental): Gross tumor volume = tumor visible on CT (+/- PET) No CTV margin will be added (Clinical target volume (CTV) = Gross target volume (GTV)) Planning Target Volume (PTV): GTV plus margins of 3-5mm (varying depending on site, motion, SABR delivery approach)
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Procedure: Minimally invasive pulmonary metastasectomy — Surgical margin is equal to tumor size, if possible The goal is a parenchymal-sparing resection
  Other Names: Lung metastasectomy
  Arms: Minimally invasive pulmonary metastasectomy
Radiation: Stereotactic ablative radiotherapy — Depending on tumor location, 54 Gy in 3 fractions, 55 Gy in 5 fractions, 60 Gy in 8 fractions.
  Other Names: SABR; Stereotactic body radiation therapy (SBRT)
  Arms: Stereotactic ablative radiotherapy

SUMMARY:
COPPER is an international, multicenter, parallel-arm, phase III randomized controlled trial comparing two local treatment strategies (SABR or metastasectomy) for patients with an indication for local treatment for limited (max. three) colorectal pulmonary metastases

DETAILED DESCRIPTION:
The study is formally endorsed by the Dutch Society of Lung Surgery (NVvL), the Dutch Society of Cardiothoracic Surgery (NVT), the Dutch Society of Radiation Oncology (NVRO). The main objective of the proposed randomized trial is to compare efficacy of SABR to the efficacy of metastasectomy with regards to the primary endpoint (local recurrence free survival at 5 years) in patients with limited colorectal pulmonary metastases. This will determine the most effective local treatment modality. The investigators hypothesize that patients with limited colorectal pulmonary metastases will have non-inferior overall survival after pulmonary metastasectomy compared to SABR, however metastasectomy will result in superior local recurrence free survival at five years when compared to SABR. In addition, the investigators hypothesize that SABR is associated with lower morbidity, comparable quality of life and comparable health care costs compared to metastasectomy. Recurrent metastases are preferably treated by the index treatment to which the patient was randomized, local recurrent metastases are preferably treated by means of cross-over between both arms. Comparing metastasectomy to SABR for patients with colorectal pulmonary metastases will present the international community the evidence needed to better select patients for local radical treatment, while diminishing uncertainty for patients and care givers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG)-Performance status 0 - 2
* Willing to provide informed consent
* Patients with 1 to 3 lung metastases from colorectal cancer eligible for both a minimally invasive surgical resection and SABR, as assessed by the multidisciplinary tumor board (MDT)
* Radically treated primary colorectal cancer
* Patient is able and willing to complete the quality-of-life questionnaires
* Previous liver metastases are radically treated with curative intent
* Histologically confirmed malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.

Exclusion Criteria:

* Previous or present metastases outside liver or lungs
* Concurrent malignant cancer, or history of other malignant cancers within the past 5 years (excluding prespecified low-risk cancers)
* Hilar or mediastinal lymph node metastases
* Poor cardiopulmonary function test
* Inability to treat all colorectal metastases
* Surgical resection by means of a bilobectomy or pneumonectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Local recurrence-free survival | From date of randomization through study completion, up to 10 years
  Time from randomization to local recurrence or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Time from randomization to death from any cause
Progression-free survival (PFS) | 5 years
  Time from randomization to disease progression at any site or death
Local recurrence rate (LRR) per tumor | 5 years
  Proportion of treated metastases with local recurrence
Quality of life (QoL) assessment - EuroQoL (EQ-5D-5L) | 5 years
  [0-5 for 5 dimensions, higher score = worse QoL]
Quality of life assessment - Functional Assessment of Cancer Therapy: General (FACT-G) | 5 years
  [27 questions in 4 subscales, higher score = better QoL]
Health economic evaluation - Institute for Medical Technology Assessment (iMTA) - iMTA Medical Cost Questionnaire (iMCQ) | 5 years
  Medical costs [Euro]
Health economic evaluation - iMTA Productivity Cost Questionnaire (iPCQ) | 5 years
  Productivity costs [Euro]
Tumor patterns of failure | 5 years
  Local, regional and distant disease control based on surveillance imaging
Rate of adverse events | 2 years
  Frequency of adverse events and serious adverse events
Multiparameter flow cytometric analyses (FACS) | 1 months
  Peripheral blood mononuclear cell (PBMC) concentration

CONTACTS AND LOCATIONS:
Overall Officials: Martijn van Dorp, MD, Principal Investigator — AUMC
Locations (1):
- Amsterdam University Medical Center (AUMC), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will become available for non-commercial scientific research (open access) after a period of 12 months after the last data collection.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Digital data and documentation will be preserved for 15 years.
Access Criteria: Data request can be done by contacting the PI.

REFERENCES:
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- [Background] Palma DA, Salama JK, Lo SS, Senan S, Treasure T, Govindan R, Weichselbaum R. The oligometastatic state - separating truth from wishful thinking. Nat Rev Clin Oncol. 2014 Sep;11(9):549-57. doi: 10.1038/nrclinonc.2014.96. Epub 2014 Jun 24. PMID 24958182
- [Background] Ritter TA, Matuszak M, Chetty IJ, Mayo CS, Wu J, Iyengar P, Weldon M, Robinson C, Xiao Y, Timmerman RD. Application of Critical Volume-Dose Constraints for Stereotactic Body Radiation Therapy in NRG Radiation Therapy Trials. Int J Radiat Oncol Biol Phys. 2017 May 1;98(1):34-36. doi: 10.1016/j.ijrobp.2017.01.204. No abstract available. PMID 28587050
- [Background] Devlin NJ, Krabbe PF. The development of new research methods for the valuation of EQ-5D-5L. Eur J Health Econ. 2013 Jul;14 Suppl 1(Suppl 1):S1-3. doi: 10.1007/s10198-013-0502-3. No abstract available. PMID 23900659
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754
- [Background] Treasure T, Farewell V, Macbeth F, Monson K, Williams NR, Brew-Graves C, Lees B, Grigg O, Fallowfield L; PulMiCC Trial Group. Pulmonary Metastasectomy versus Continued Active Monitoring in Colorectal Cancer (PulMiCC): a multicentre randomised clinical trial. Trials. 2019 Dec 12;20(1):718. doi: 10.1186/s13063-019-3837-y. PMID 31831062
- [Background] Lodeweges JE, Klinkenberg TJ, Ubbels JF, Groen HJM, Langendijk JA, Widder J. Long-term Outcome of Surgery or Stereotactic Radiotherapy for Lung Oligometastases. J Thorac Oncol. 2017 Sep;12(9):1442-1445. doi: 10.1016/j.jtho.2017.05.015. Epub 2017 May 30. PMID 28576747
- [Background] Nelson DB, Tayob N, Nguyen QN, Erasmus J, Mitchell KG, Hofstetter WL, Sepesi B, Antonoff MB, Mehran RJ. Local failure after stereotactic body radiation therapy or wedge resection for colorectal pulmonary metastases. J Thorac Cardiovasc Surg. 2019 Oct;158(4):1234-1241.e16. doi: 10.1016/j.jtcvs.2019.02.133. Epub 2019 May 11. PMID 31395367
- [Background] van Dorp M, Gonzalez M, Daddi N, Batirel HF, Brunelli A, Schreurs WH. Metastasectomy for colorectal pulmonary metastases: a survey among members of the European Society of Thoracic Surgeons. Interdiscip Cardiovasc Thorac Surg. 2023 Feb 6;36(2):ivad002. doi: 10.1093/icvts/ivad002. PMID 36847670
- [Background] Nicosia L, Franceschini D, Perrone-Congedi F, Casamassima F, Gerardi MA, Rigo M, Mazzola R, Perna M, Scotti V, Fodor A, Iurato A, Pasqualetti F, Gadducci G, Chiesa S, Niespolo RM, Bruni A, Alicino G, Frassinelli L, Borghetti P, Di Marzo A, Ravasio A, De Bari B, Sepulcri M, Aiello D, Mortellaro G, Sangalli C, Franceschini M, Montesi G, Aquilanti FM, Lunardi G, Valdagni R, Fazio I, Scarzello G, Corti L, Vavassori V, Maranzano E, Magrini SM, Arcangeli S, Gambacorta MA, Valentini V, Paiar F, Ramella S, Di Muzio NG, Livi L, Jereczek-Fossa BA, Osti MF, Scorsetti M, Alongi F. A multicenter LArge retrospectIve daTabase on the personalization of stereotactic ABlative radiotherapy use in lung metastases from colon-rectal cancer: The LaIT-SABR study. Radiother Oncol. 2022 Jan;166:92-99. doi: 10.1016/j.radonc.2021.10.023. Epub 2021 Nov 5. PMID 34748855
- [Background] Franks KN, McParland L, Webster J, Baldwin DR, Sebag-Montefiore D, Evison M, Booton R, Faivre-Finn C, Naidu B, Ferguson J, Peedell C, Callister MEJ, Kennedy M, Hewison J, Bestall J, Gregory WM, Hall P, Collinson F, Olivier C, Naylor R, Bell S, Allen P, Sloss A, Snee M. SABRTooth: a randomised controlled feasibility study of stereotactic ablative radiotherapy (SABR) with surgery in patients with peripheral stage I nonsmall cell lung cancer considered to be at higher risk of complications from surgical resection. Eur Respir J. 2020 Nov 12;56(5):2000118. doi: 10.1183/13993003.00118-2020. Print 2020 Nov. PMID 32616595